CLINICAL TRIAL: NCT06665698
Title: Prospective Study to the Evaluate the Long-term Use of Synthetic I-STOP® Device for Treatment of Stress Urinary Incontinence in Women
Brief Title: Long-term Evaluation of the I-STOP Sling in Stress Urinary Incontinence Treatment
Acronym: VIGI-ISTOP
Status: Not yet recruiting | Type: Observational
Sponsor: DILO Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: VI-IS-24
Record Dates: First submitted 2024-10-25; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: I-STOP; MUS; Sling
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Evaluate quality of life and rate of reoperation after implantation of the I-STOP sling for stress urinary incontinence

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-comparative, interventional post-marketing clinical follow-up study (PMCF) on a population of patients with SUI requiring surgical treatment with implantation of an I-STOP sling to document safety, the performance and effectiveness in the short, medium, and long term of these I-STOP® implants used in their intended purpose.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman aged over 18 ;
* Patient with SUI, having escaped "conservative" medical treatment, with indication for surgical treatment with implantation of an I-STOP® strip via trans-obturator or retropubic route as indicated in the instructions for use of the SUI implant ;
* Patient affiliated to a social security scheme;
* Patient capable of completing a self-questionnaire;
* Patient able to understand the protocol and follow the visit schedule;
* Patient having signed informed consent.

Exclusion Criteria:

* Minor patient, pregnant or breastfeeding ;
* Adult patient subject to a measure of legal protection, guardianship, curatorship or deprived of liberty by judicial or administrative decision ;
* Patient presenting a contraindication to the use of the implant indicated in the instructions for use of the implant ;
* Patient with a medical contraindication to surgery and/or anaesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is made up of patients with SUI who should benefit from the implantation of an I-STOP® implant in one of the centers associated with the project.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Rate of reintervention | One year after surgery and after each year during 10 years
  Questionnaire sent every year to the patient with question about revision surgery: yes / no

SECONDARY OUTCOMES:
Quality of Life | One year after surgery and after each year during 10 years
  Questionnaire sent every year: Pelvic Floor Impact Questionnaire-short form 7 (PFIQ-7)

IPD SHARING:
Plan to Share IPD: Undecided